CLINICAL TRIAL: NCT01771874
Title: Influence of Bupropion on the Effects of MDMA
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: University Hospital, Basel, Switzerland (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: Quadruple | Purpose: Basic Science
Other Study IDs: EK 190/12
Record Dates: First submitted 2012-10-24; First posted 2013-01-18 (Estimated); Last update posted 2016-01-21 (Estimated); Status verified 2016-01

CONDITIONS: Healthy; Substance-related Disorders
Keywords: MDMA; pharmacokinetics; pharmacodynamics; emotions; Mechanism of action of MDMA; Interaction study; Effect of MDMA and bupropion on emotions
MeSH Terms: conditions — Substance-Related Disorders | interventions — N-Methyl-3,4-methylenedioxyamphetamine; Bupropion

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- MDMA, bupropion, placebo (Experimental): Cross-over within-subjects design with all treatment conditions tested in the same subject. This design has 1 arm but two (actually 4) treatment conditions in the same subject. The four treatment conditions are placebo-placebo, bupropion-placebo, placebo-MDMA, and bupropion-MDMA.
  Interventions: Drug: MDMA; Drug: Bupropion; Drug: Placebo

INTERVENTIONS:
Drug: MDMA — 125 mg per os, single dose
  Other Names: Ecstasy; 3,4-Methylenedioxymethamphetamine
Drug: Bupropion — Bupropion will be administered in a dose of 150mg (Wellbutrin XR) once-daily in the morning for three days followed by 300mg (2x150mg) for 4 days before the test day. On the test day, a final dose of 300mg will administered 2 hours before the administration of MDMA 125 mg or placebo.
  Other Names: Wellbutrin XR; Zyban
Drug: Placebo — per os
  Other Names: capsules containing manitol looking identical to MDMA or bupropion

SUMMARY:
The purpose of this study is to determinate the effect of a pre-treatment with bupropion, a dopamine and norepinephrine transporter inhibitor, on the pharmacodynamics and pharmacokinetics of 3,4-methylenedioxymethamphetamine (MDMA, "Ecstasy"). The study will provide further understanding of the dopaminergic regulation of mood.

DETAILED DESCRIPTION:
3,4-methylenedioxymethamphetamine (MDMA, "ecstasy") is widely used by young people for its euphoric effects. MDMA releases serotonin (5-HT), dopamine (DA), and norepinephrine (NE). 5-HT release mainly contributes to the subjective effects of MDMA whereas NE release is involved in the cardiovascular and psychostimulant effects of MDMA. DA mediates the reinforcing addiction-related effects of drugs of abuse but it is unclear whether DA contributes to the acute effects of MDMA in humans. To determine the role of DA transporter-mediated DA release in the acute response to MDMA in humans the investigators test the effects of the DA transporter inhibitor bupropion on the physiological and subjective effects of MDMA. The investigators use a randomized double-blind placebo-controlled cross-over design with four experimental sessions. Bupropion or placebo will be administered before MDMA or placebo to 16 healthy volunteers. Subjective and cardiovascular responses will be repeatedly assessed throughout the experiments and plasma samples are collected for pharmacokinetics. The primary hypothesis is that bupropion reduces the MDMA-induced increase in positive mood.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 and 45
* Understanding of the German language
* Subjects understand the procedures and the risks associated with the study
* Participants must be willing to adhere to the protocol and sign the consent form
* Participants must be willing to adhere to the protocol and sign the consent form
* Participants must be willing to drink only alcohol-free liquids and no xanthine-containing products(such as coffee, black or green tea, red bull, chocolate) after midnight of the evening before the study session, as well as during the study day
* Participants must be willing not to drive a traffic vehicle within 48 h following MDMA administration
* Women of childbearing potential must have a negative pregnancy test at the beginning of the study and must agree to use an effective form of birth control. Pregnancy tests are repeated before each study session
* Body mass index: 18-27 kg/m2

Exclusion Criteria:

* Chronic or acute medical condition including clinically relevant abnormality in physical exam, laboratory values, or ECG. In particular: Hypertension (>140/90 mmHg) or Hypotension (SBP<85 mmHg). Personal or first-grade history of seizures. Cardiac or neurological disorder
* Current or previous psychotic or major affective disorder
* Psychotic or major affective disorder in first-degree relatives
* Prior illicit drug use (except tetrahydrocannabinol (THC)-containing products) more than 5 times or any time within the previous 2 months
* Pregnant or nursing women
* Participation in another clinical trial (currently or within the last 30 days)
* Use of medications that are contraindicated or otherwise interfere with the effects of the study medications (monoamine oxidase inhibitors, antidepressants, sedatives etc.)
* Tobacco smoking

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 16 (Actual)
Dates: Start 2013-01; Primary Completion 2013-05 (Actual); Study Completion 2013-09 (Actual)

PRIMARY OUTCOMES:
Positive Mood Effects | 24 hours
  A significant reduction of the (100-mm Visual Analog Scale) positive mood response to MDMA by bupropion.

SECONDARY OUTCOMES:
Blood pressure(mmHg)during 10 hours | 10 hours
Neuroendocrine plasma levels | 10 hours
  assessed: prolactin, cortisol, epinephrine, norepinephrine, oxytocin, pro-vasopressin, vasopressin, estrogen,and progesterone
Drug plasma levels | 24 hours
  The plasma concentration of MDMA and bupropion is repetitively assessed
Heart rate (bpm) | 10 hours
Body temperature | 10 hours
Effects on social cognition (emotion recognition and empathy) | 10 hours
Influence of genetic cytochrome P450 2D6 polymorphisms on the metabolism of MDMA | 24hours
  We will assess the effects of the subjects' genotype and phenotype on MDMA and its metabolites plasma concentrations.

CONTACTS AND LOCATIONS:
Overall Officials: Matthias E Liechti, MD, MAS, Principal Investigator — University Hospital, Basel, Switzerland
Locations (1):
- University Hospital Basel, Basel, Canton of Basel-City, Switzerland

REFERENCES:
- [Derived] Vizeli P, Liechti ME. Oxytocin receptor gene variations and socio-emotional effects of MDMA: A pooled analysis of controlled studies in healthy subjects. PLoS One. 2018 Jun 18;13(6):e0199384. doi: 10.1371/journal.pone.0199384. eCollection 2018. PMID 29912955
- [Derived] Boxler MI, Liechti ME, Schmid Y, Kraemer T, Steuer AE. First Time View on Human Metabolome Changes after a Single Intake of 3,4-Methylenedioxymethamphetamine in Healthy Placebo-Controlled Subjects. J Proteome Res. 2017 Sep 1;16(9):3310-3320. doi: 10.1021/acs.jproteome.7b00294. Epub 2017 Aug 9. PMID 28722422